CLINICAL TRIAL: NCT01292902
Title: Regional Distribution of Ventilation in Patients With Chronic Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Armèle de Fátima Dornelas de Andrade, Universidade Federal de Pernambuco
Model: Parallel | Masking: None
Other Study IDs: 27012011
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Last update posted 2011-02-10 (Estimated); Status verified 2011-01

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- healthy volunteers (Active Comparator)
  Interventions: Other: inspiratory muscle exercise
- chronic heart failure (Other)
  Interventions: Other: inspiratory muscle exercise

INTERVENTIONS:
Other: inspiratory muscle exercise — To conduct the exercise to the inspiratory muscles was used for IMT Threshold ® device (Threshold Inspiratory Muscle Trainer, HealthScan Products Inc., Cedar Grove, New Jersey) is one of the most used for training of inspiratory muscles in patients with several pathologies such as ICC.Threshold ® has been engaged in the patient's mouth by a mouthpiece, with the nose occluded by a nose clip. The exercise time was 3 minutes. During this period, participants were encouraged to only breathe through the mouth and maintain a respiratory rate between 12 and 16ipm. The exercise would be stopped if HR increased more than 20% and / or SpO2 < 88%.
  Arms: chronic heart failure
Other: inspiratory muscle exercise — Equal to the group with chronic heart failure.
  Arms: healthy volunteers

SUMMARY:
Inspiratory muscle dysfunction is a reduction in the ability to generate pressure and force by the inspiratory muscles. This decrease in the strength of these muscles can be attributed to biochemical and histological changes. Some patients with CHF showed a reduction of maximal inspiratory pressure (MIP) and inspiratory muscle endurance, and such factors known to exercise limitation and deterioration in quality of life and worsens the prognosis of these patients. This study aims to evaluate the Regional pulmonary distribution volume and the influence of enclosures system thoracoabdominal in CHF patients with cardiomegaly associated with diaphragmatic weakness during quiet breathing and during exercise for inspiratory muscle and its correlation with functional data. The investigators evaluated a total of 31 individuals divided into two groups: CHF and control. In the control group, twelve volunteers participated with similar age, gender and body mass index in relation to the group of patients with CHF. The control group participants had an ejection fraction of left ventricle (EF)> 50% without cardiac abnormalities of the cameras and MIP over 80% of predicted. To conduct the exercise to the inspiratory muscles (EMI) was used for IMT Threshold ® device (Threshold Inspiratory Muscle Trainer, HealthScan Products Inc., Cedar Grove, New Jersey) is one of the most used for training of inspiratory muscles in patients with several pathologies such as CHF. The exercise time was 3 minutes. During this period, participants were encouraged to only breathe through the mouth and maintain a respiratory rate between 12 and 16ipm. Opto-electronic plethysmography measures the volume changes of thoracoabdominal system by placing 89 markers formed by hemiesferas covered with retro-reflective paper, taking the place of each of these hemiesferas determined by anatomical landmarks on the anterior and posterior regions of the chest and abdomen. According to our study, a lower ventilation on diaphragmatic region would lead to an increased perception of dyspnea during submaximal exercise in this population. Moreover, the observed changes in the pattern of regional distribution of ventilation in CHF patients compared to healthy individuals can serve as a basis for prospective cohort studies using IMT.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as CHF associated with cardiomegaly
* Class II and III (NYHA)
* Left ventricular minor 45% (method Teicholtz)
* Inspiratory muscle weakness (PiMáxima <70% predicted)
* Duration of symptoms > 1 year
* Body mass index (BMI) < 35kg/m2
* Non-smokers or former smokers with a smoking history < 10 pack-years

Exclusion Criteria:

* Patients with chronic heart failure who had unstable angina, myocardial infarction or heart surgery until three months before the survey
* Orthopedic diseases or respiratory comorbidities such as asthma and COPD

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Opto-electronic plethysmography | 1 year
  The POE (BTS Bioengineering, Italy) measures the volume changes of thoracoabdominal system through placement of 89 markers formed by hemiesferas covered with retro-reflective paper, taking the place of each of these hemiesferas determined by anatomical landmarks in anterior and posterior thorax and abdomen.

SECONDARY OUTCOMES:
Assessment of Functional Capacity | 1 year
  To assess the functional capacity test was used for 6-minute walk (6MWT) according to the protocol established by the American Thoracic Society (ATS). Before the test parameters were assessed resting blood pressure (BP), Heart Rate (HR), Oxygen Saturation (SpO2 - pulse oximetry portable Onix 9500), Respiratory Frequency (RF) and dyspnea scale (scale Borg).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Pernamabuco, Recife, Pernambuco, Brazil

REFERENCES:
- [Result] Ernst ER, Shub C, Bailey KR, Brown LR, Redfield MM. Radiographic measurements of cardiac size as predictors of outcome in patients with dilated cardiomyopathy. J Card Fail. 2001 Mar;7(1):13-20. doi: 10.1054/jcaf.2001.23244. PMID 11264545